CLINICAL TRIAL: NCT03457792
Title: Abatacept in Early-Stage Rheumatoid Arthritis Patients: Longterm Experience and Efficacy in Routine Clinical Practice
Brief Title: A Study of Abatacept in Participants That Only Recently Started to Develop Rheumatoid Arthritis
Acronym: ASCEND
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-679
Record Dates: First submitted 2018-02-13; First posted 2018-03-08 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Abatacept for Rheumatoid Arthritis (RA): Participants diagnosed with moderate to severe active RA within the last 24 months and initiated treatment with Abatacept

SUMMARY:
This is a long-term study of Abatacept in participants that only recently started to develop Rheumatoid Arthritis, a chronic inflammatory disorder affecting mainly joints.

ELIGIBILITY:
Inclusion Criteria:

* Participants recently (within the last 24 months before enrollment) diagnosed with established moderate to severe active RA
* Participants naïve of abatacept and who, at their physician's discretion, are initiated with abatacept according the German label/SmPC (Summary of product characteristics)

Exclusion Criteria:

* Participants who are currently included in any interventional clinical trial in RA

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participant population targeted in this study consists of participants with early-stage RA (i.e. diagnosis of RA not longer than 24 months) that initiate treatment with Abatacept.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Number of patients continuing with abatacept treatment | Up to 12 months

SECONDARY OUTCOMES:
Anti-citrullinated protein antibody (ACPA) titer | At baseline
Concomitant treatment given with abatacept as determined by the investigator | Up to 12 months
Dosage of abatacept as determined by the investigator | Up to 12 months
Frequency of administration of abatacept | Up to 12 months
Reason for abatacept treatment initiation as determined by the investigator | At baseline
Number of patients previously receiving disease modifying anti-rheumatic drug (DMARD) | Up to 12 months
Socio-demographics of participants as determined by the investigator | At baseline
Disease history of participants as determined by the investigator | At baseline
Number of patients with cardiovascular risk factors (smoker, hypertension, diabetes, dyslipidemia) | Up to 12 months
Number of patients with other pathologies (cardiovascular, respiratory, liver, renal, cancer, infections, and immuno-deficiency) | Up to 12 months
Simplified Disease Activity Score (based on 28 joints) (DAS28) | Up to 12 months
  DAS28: Swollen joint count [SJC], tender joint count [TJC], C-reactive protein [CRP], erythrocyte sedimentation rate [ESR]
Number of patients who achieve the first response to treatment per European League Against Rheumatism (EULAR) response criteria | Up to 12 months
Number of patients who achieve the first clinically significant Disease Activity Score (DAS)-change (≥ 1.2) | Up to 12 months
Number of patients who achieve the first low disease activity score (LDAS), DAS28 ≤ 3.2 | Up to 12 months
Number of patients who achieve the first remission state, DAS28 < 2.6 | Up to 12 months
Number of Adverse Events (AE) | Up to 12 months
Number of Serious Adverse Events (SAE) | Up to 12 months
Health Assessment Questionnaire Disability Index (HAQ-DI) | Up to 12 months
Existence or the absence of radiographic erosions as determined by the investigator by imaging technique | At baseline
Existence or the absence of radiographic erosions as determined by the investigator by imaging technique | Up to 12 months
Rheumatoid factor (RF) | Up to 12 months
Patient global assessment (PGA) | Up to 12 months
Evaluator global assessment (EGA) | Up to 12 months
Clinical disease activity index (CDAI) | Up to 12 months
Simple disease activity index (SDAI) | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Freiburg im Breisgau, Germany

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome